CLINICAL TRIAL: NCT03735953
Title: Retroflexion in the Entire Colon for the Detection of Colon-related Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 20181030
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Colon Cancer Screening; Colon Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retroflexion arm (Experimental): Retroflexion in the total colon and slow withdrawal to the rectum and record all visible colon polyps and other colon related diseases
  Interventions: Diagnostic Test: Retroflexion in the total colon
- Forward view arm (No Intervention): Colonoscope is slowly withdrawn from the proximal colon to the the rectum have a forward view and record all visible colon polyps and other colon related diseases

INTERVENTIONS:
Diagnostic Test: Retroflexion in the total colon — retroflexion in the cecum or proximal ascending colon and slow withdrawal to the rectum
  Arms: Retroflexion arm

SUMMARY:
Colorectal cancer is one of the common gastrointestinal malignancies, and the incidence of colorectal cancer in China increases by 3% to 4% annually . Colorectal adenoma is the most important precancerous lesion of colorectal cancer. Timely screening for colorectal adenoma and endoscopic resection is the most effective measure to prevent colorectal cancer .Removal of pre-malignant colon polyps during colonoscopy reduces colorectal cancer mortality by over 50%. However,Conventional colonoscopy endoscopy is a direct-view type, and the visual field is limited. About 10%-24% of the lesions may be missed. The ascending colon is more difficult because of the deep folds, and the rate of missed diagnosis is higher. Our goal is to determine if additional pre-cancerous colon polyps can be identified by looking at the total colon in retroflexion. During retroflexion the tip of the colonoscope is turned 180 degrees; allowing the doctor to view the backs of colonic folds. If additional polyps can be identified in this manner colonoscopy will become a more efficient method of screening for colon cancer.

In order to evaluate how effective colon retroflexion is at detecting polyps in the total colon the investigators plan on performing a randomized, controlled trial. Patients undergoing screening or follow up colonoscopy will be invited to participate in the study. Those patients who agree to participate will be randomized into one of two groups once the colonoscope is fully inserted. Group one will have their colon examined for polyps with the endoscope looking forward (traditional form of examination) followed by repeat examination of the total colon with the colonoscope in retroflexion (looking backwards). In group two the colonoscopy will be completed in the usual manner. Polyps seen during each section of the exam will be recorded. The duration of each portion of colonoscopy will be recorded. After the procedure is completed the physician performing the colonoscopy will rate difficulty of the procedure and confidence with quality of the examination. Assess and record the degree of pain during and after the patient's examination.Pathology results for each polyp will be recorded once available. There will be no study related follow up after the pathology results are recorded.

DETAILED DESCRIPTION:
Colorectal cancer is one of the common malignant tumors of the digestive tract. The incidence of colorectal cancer in China has increased by 3%-4% annually . Colorectal adenoma is the most precancerous lesion of colorectal cancer. Screening for colorectal adenoma and endoscopic resection are the most effective measures to prevent colorectal cancer . Colonoscopy and endoscopic polypectomy can effectively prevent the occurrence of colorectal cancer, and it can reduce the mortality of colorectal cancer by more than 50% . Especially in the rectum and sigmoid colon and other high-intestinal segments of colorectal cancer, the reduction effect is very significant . However, colonoscopy, currently considered a "gold standard," still misses a significant number of lesions. A foreign meta-analysis showed that the rate of missed diagnosis of polyps in colonoscopy was as high as 22% . Especially for the right colon, the protective effect of colonoscopy is not ideal, and the incidence of right inter-coloanal cancer is significantly higher than that of the left colon . This difference may be caused by tumorigenesis and polyp morphology in the right colon and left colon. Flat polyps, which are more common in the right colon, are more likely to be missed than pedicle polyps, which are more common in the left colon. In addition, it is more difficult to observe the polyps in the right colon fold by conventional colonoscopy. Over the years, techniques to improve the positive rate of diagnosis of the right Semi-colon have emerged, including providing high-quality bowel preparation, setting up a standard time for the right Semi-colon independent decolonisation, repeated screening of the right Semi-colon and the conduct of the ascending colon inversion .

Inversion technique is a special method of examination in colonoscopy. It was first used by Grobe in the examination of rectal lesions in 1982 and achieved good results. In addition, for some polyps near the proximal rectum, which are difficult to reach with endoscopy, the application of this technique can effectively perform polypectomy . At present, the most popular in the lower digestive tract examination is the inversion technique of the rectal abdomen, but it has not been popularized in colon examination . Conventional colonoscopy endoscopy is a direct-view type, and the visual field is limited. About 10%-24% of the lesions may be missed. The ascending colon is more difficult because of the deep folds, and the rate of missed diagnosis is higher. The colon reversal technique can observe the oral mucosa of the colonic meniscus, increase the observation of the colonic mucosa, and make up for the defects of the conventional retrospective, which is crucial for improving the positive rate of colonic lesion diagnosis. During retroflexion the tip of the colonoscope is turned 180 degrees; allowing the doctor to view the backs of colonic folds. If additional polyps can be identified in this manner colonoscopy will become a more efficient method of screening for colon cancer.However, inversion techniques may increase the incidence of complications and increase the time of examination to bring some painful experience to the subject. At present, there are many endoscopic reversal studies on the right colon in China and abroad. Luo Yuanqiang and Chen Peisong and other studies have found that ascending colonic reversal can improve the detection rate of polyposis and reduce the rate of polyps missed .A foreign meta-analysis showed that the inversion technique of the right colon can significantly increase the rate of adenoma discovery without increasing the incidence of adverse events . However, there is no research on total colon reversal at domestic and abroad. Observation of reversal of the whole colon may increase the detection rate of related lesions, but it may also increase the examination time and adverse events, and because colonoscopy has a relatively high rate of detection of left colonic lesions, so the investigators need to fully evaluate the overall colon inversion technique for disease detection rate and the degree of pain and adverse events in the subject.

This study aimed to evaluate the value of inversion techniques in improving the detection rate of colorectal polyps and its safety and operational feasibility by comparing the inversion method with conventional direct observation method by randomized controlled method.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age undergoing colonoscopy for colorectal cancer screening or routine polyp surveillance

Exclusion Criteria:

* Failure to intubate the cecum during colonoscope insertion
* Prior right colon resection
* Known polyposis syndrome or polyposis identified at colonoscopy
* Inflammatory bowel disease
* Preparation of the colon is judged fair or poor using Boston Bowel Preparation Scale.
* Severe cardio-cerebral diseases
* Pregnant women, lactating women
* Acute lower gastrointestinal bleeding
* Preoperative use of antispasmodic sedative drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-11-20 (Estimated)

PRIMARY OUTCOMES:
per-patient adenoma and polyp detection rate | 1 day
  Patients were randomized to the exam of the proximal colon in forward or retroflexion view , and adenoma detection rates compared.

SECONDARY OUTCOMES:
Total procedure time | 1 day
  Total procedure time including intubation and withdrawal time
Rate of retroflexion-related adverse events. | through study completion, an average of 1 year
  Rate of retroflexion-related adverse events.
Patient's feeling | In colonoscopy, at the end of the examination and 1 hour, 6 hours, 12 hours after the examination
  patients' feeling, quantified using visual analogue scale from 0 (no pain) to 10 (severe pain that is unbearable.)

CONTACTS AND LOCATIONS:
Overall Officials: Baicang Zou, MD, Study Director — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohen J, Grunwald D, Grossberg LB, Sawhney MS. The Effect of Right Colon Retroflexion on Adenoma Detection: A Systematic Review and Meta-analysis. J Clin Gastroenterol. 2017 Oct;51(9):818-824. doi: 10.1097/MCG.0000000000000695. PMID 27683963
- [Result] Kushnir VM, Oh YS, Hollander T, Chen CH, Sayuk GS, Davidson N, Mullady D, Murad FM, Sharabash NM, Ruettgers E, Dassopoulos T, Easler JJ, Gyawali CP, Edmundowicz SA, Early DS. Impact of retroflexion vs. second forward view examination of the right colon on adenoma detection: a comparison study. Am J Gastroenterol. 2015 Mar;110(3):415-22. doi: 10.1038/ajg.2015.21. Epub 2015 Mar 3. PMID 25732415